CLINICAL TRIAL: NCT05637723
Title: Evaluation of the Efficacy of Three-Dimensional Schroth Exercises on Pelvic Asymmetry and Pelvic Floor Muscles in Patients With Adolescent Idiopathic Scoliosis
Brief Title: The Effect of Schroth Exercises on Pelvic Floor Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep Ayyıldız Eroğlu, MSc Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schroth Exercise
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Scoliosis
Keywords: scoliosis; pelvic floor muscle; schroth exercise
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- schroth exercise group (Experimental): Included participants will be included in the Schroth exercise program by a Schroth-trained physiotherapist 3 days a week for 6 weeks, after being evaluated at the start of treatment.
  Interventions: Other: schroth exercise
- traditional scoliosis exercise group (Active Comparator): Included participants will be included in the traditional scoliosis exercise program by a physiotherapist 3 days a week for 6 weeks, after being evaluated at the start of treatment.
  Interventions: Other: traditional scoliosis exercises
- control group (No Intervention): Any exercise program for scoliosis will not be applied to this group.

INTERVENTIONS:
Other: schroth exercise — The schroth exercise program will be given 3 days a week for 6 weeks.
  Arms: schroth exercise group
Other: traditional scoliosis exercises — The traditional scoliosis exercises program will be given 3 days a week for 6 weeks.
  Arms: traditional scoliosis exercise group

SUMMARY:
The aim of this study is to evaluate the effect of Schroth exercise training and Traditional Scoliosis exercise training applied 3 days a week for 6 weeks in people with Adolescent Idiopathic Scoliosis on the pelvic floor muscles and to compare these results with the control group, to evaluate pelvic asymmetry, pain, posture, body awareness, flexibility and life expectancy. It will be planned as a prospective randomized controlled trial to evaluate the correlation between 3 groups on the quality of life.

DETAILED DESCRIPTION:
Scoliosis is defined as the lateral curvature of the spine more than 10 degrees to the right or left, detected radiologically in the coronal plane, but scoliosis is a complex three-dimensional orthopedic deformity that also affects the spine, shoulder girdle and pelvis. The etiopathogenesis of scoliosis is still unclear and the cause cannot be determined in 80% of cases, and it is called idiopathic scoliosis. Other causes include neurological, bone origin, trauma, joint and connective tissue pathologies. Scoliosis causes postural changes in the whole body of the person due to the rotation and angulation of the spine. Especially the abdominal muscles, rib cage, back and waist extensors are most affected by this condition, and it causes biomechanical changes in the pelvis, shoulder girdle and even lower extremities and feet. The spine causes severe morphological changes due to vertebral wedging and rib cage distortion. Vertebral wedging causes a progressive vertebral deformation associated with axial rotation and scoliosis progression. This vertebral deformation is not only associated with the deterioration of the bone structure and the spine, but also causes changes in the structures of the upper extremity and lower extremity. In the treatment of scoliosis; There are four main categories as observation, corset, physiotherapy and rehabilitation applications and surgery. These treatments should be decided by considering the risk of curvature progression. The main purpose in the treatment of scoliosis is to prevent curvature progression. In scoliosis, besides the spine, the shoulder girdle, pelvis and even the lower extremities are also affected by this pathological condition and postural problems occur. Therefore, a detailed clinical analysis and evaluation of the entire musculoskeletal system should be performed in individuals with scoliosis. The problem is determined by revealing in detail the length, strength and functional status of the muscles and ligaments that cause impaired body cosmetics. It has been reported in the literature that pelvic anomalies occur with the progression of scoliosis. Qui et al. reported that there is a difference between the right and left of the pelvis, which is not due to developmental asymmetry or distortion of the pelvis, but due to horizontal rotation. At the same time, Gum et al. reported that people with adolescent idiopathic scoliosis (AIS) have advanced pelvic rotations in the transverse plane. Stylianides et al. reported for the first time iliac crest asymmetry in people with untreated AIS using 3D electromagnetic pointers. In individuals with severe scoliosis angles, skeletal deformity of the spine is associated with pelvis misalignment and morphological asymmetry. The importance of spinopelvic parameters has been reported when defining sagittal balance in scoliosis. The European Society of Scoliosis Orthopedics and Rehabilitation (SOSORT) recommends scoliosis-specific exercises in addition to bracing for scoliosis. It has been reported that the progression of the curve is very rapid if there is a progression of 5.4 degrees and above in the measurements taken every 6 months for curves of 25 degrees and above and these people should be included in the treatment. Although bracing is a difficult treatment to accept in some children, the acceptance of exercise therapy is higher. Schroth exercises are specialized exercises for scoliosis and have been reported to reduce the Cobb angle of curvature, improve neuromotor control, increase respiratory function and back flexibility, and improve cosmetic appearance. The Schroth method includes scoliosis-specific sensorimotor, posture and breathing exercises, and provides the prevention of 3-dimensional spinal deformities in the spine by the formation of postural realignment in people with AIS. With the autocorrection included in the method, self-elongation and postural correction are provided to each curvature pattern and the person's muscle imbalance is balanced. It has been reported that with Schroth exercises, muscle strength and flexibility are increased, the Cobb angle is improved, and surgery rates are reduced. Schreiber et al. reported a significant difference in pain, curvature progression and body awareness in the intervention group in which they included 50 people with AIS, compared to the control group. In this study, in which the endurance of the back muscles was evaluated for the first time, the Schroth intervention group showed improvement. In another study by Schreiber et al., it was reported that Schroth exercises had positive effects on reducing the progression of the curvature. Although it has been reported that the strength of the back muscles is increased with schroth exercises, there is no study in the literature reporting the relationship between pelvic floor muscles and schroth exercises in individuals with scoliosis. The aim of this study is to evaluate the effectiveness of the Schroth method on pelvic floor muscle activity and pelvic asymmetry in people with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with idiopathic scoliosis by a specialist physician,
* 7-25 years old,
* The primary curvature is between 10-45 degrees according to the Cobb method,
* C or S scoliosis,
* Pain in the back/lumbar region due to scoliosis,
* Those who have not received any exercise therapy for scoliosis before,
* Volunteer to participate in the study,
* Having the cognitive capacity to cooperate with the guidance of the physiotherapist,
* Have not had any musculoskeletal injury in the last 6 months,
* No neurological, orthopedic or cardiopulmonary disorders other than the diagnosis of scoliosis,
* Young individuals who have not undergone any surgery related to the diagnosis of scoliosis will be included in the study.

Exclusion Criteria:

* The patient has any contraindications for exercise,
* Having previously undergone spine surgery and pelvic surgery,
* Having any mental problems,
* The fact that scoliosis is not idiopathic but has arisen for different reasons (neurological, congenital),
* In case of neurological, psychiatric, muscular, rheumatic or orthopedic diseases, these people will not be included in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of pelvic floor muscle strength | 6 weeks
  The ability of the pelvic floor muscles to contract and relax is evaluated by contraction and relaxation of the pubococcygeal muscles around the vagina and anus. In our study, we will try to determine the change in pelvic floor muscle activity before and after Schroth treatment using EMG Biofeedback device. EMG Biofeedback will be used for evaluation purposes.
Assessment of cobb angle | 6 weeks
  The degree of curvature in the coronal plane is measured radiographically according to the Cobb method. The Cobb angle, considered the gold standard, is the angle between the perpendiculars when descending lines drawn from the top of the curve along the upper endplate of the most tilting vertebra at the top and the lines drawn under the lower endplate of the most tilting vertebrae to the bottom. The Cobb angle describes only one plane of a three-dimensional deformity, but provides information about the progression of the curvature. Observer variability was recorded as 2.8°-4.9° and interobserver variability was recorded as 6.3°-7.2° in Cobb angle measurement with conventional techniques. In digital Cobb angle measurements, the variability for the same observer and the interobserver variability were reported as 1.3°. In the study, it is planned to evaluate the Cobb angle by the relevant physician.

SECONDARY OUTCOMES:
Assessment of Risser sign | 6 weeks
  The epiphyseal plate starts from the lateral border of the anterior superior spina iliaca, runs medially, and ends at the posterior superior spina iliaca. The degree of completion is expressed as a percentage: Grade 1 ≤ 25%, Grade 2 26-50%, Grade 3 51-75%, Grade 4 75-100%. When the epiphysis is combined with the illium, it is defined as Grade 5. The Risser sign is used to determine the age of bone development, growth rate and risk level for scoliosis. In the study, it was used to determine the age of bone development. It has been reported to be reliable and sensitive in determining the age of bone development.
Assessment of Angle of Trunk Rotation | 6 weeks
  Measurement of trunk rotation angle/degree is the most appropriate method used in the clinical evaluation of scoliosis. ATR can be used to monitor the effects of treatment without radiographic evaluation. ATR measurement is done using a special inclinometer called a scoliometer. The patient is asked to lean forward with the arms relaxed. The scoliometer is placed posteriorly and the degree observed at the point of greatest gibbosis is recorded. ATR is a reliable measurement with a repeatability of 86%. A variation of 2° in interobserver measurements can be considered significant. In this study, it is planned to evaluate ATR measurements before and after treatment with a Scoliometer® brand scoliometer. There is a correlation between the Scoliometer® and the Cobb angle. The Scoliometer® has been observed to have specificity, sensitivity and predictive ability. Intra-rater and inter-rater reliability coefficients are r = .86-.97
Assessment of trunk flexibility | 6 weeks
  In the trunk flexion flexibility test, the person will try to touch the fingertips with their hands from a standing position on a 15 cm high block without bending the knees, and the distance between the fingertip and the tatha block surface will be measured with a tape measure. Flexibility of trunk lateral flexion will be evaluated by measuring the distance between the middle finger of the right hand in the standing position and after complete lateral flexion. Each measurement will be repeated 3 times and the average of the 3 measurements will be taken.
Assessment of Posture | 6 weeks
  Posture assessment of young individuals included in the study was performed by McRoberts et al. It will be done with the New-York Posture Scale (NYPRS), which has been proven to be reliable in assessing changes in postural alignment. Evaluation with this scale is made by observing the postural changes that may occur in 13 different parts of the body. Accordingly, if the person has a correct posture, he/she gets 5 points, if the posture is moderately impaired, 3 points, and 1 point if there is a serious deterioration in posture. The maximum score obtained as a result of the test is 65, the minimum score is 13, and higher scores indicate better postural alignment. According to the standard evaluation criteria developed for this test, the posture of the person was evaluated over a total of 65 points. " and 19 will be recorded as "bad"
Assessment of Body Awareness | 6 weeks
  Body awareness of the individuals included in the study was first evaluated by Shields SA et al. Karaca S. et al. It will be evaluated by using the Turkish version with proven validity and reliability on university students. VFA consists of four subgroups (changes in body process, sleep-wake cycle, prediction of onset of illness, prediction of body responses) aiming to determine the level of normal or abnormal sensitivity to body composition and "I understand the difference in my body's responses to various foods", "I can predict I will have the flu". It is a questionnaire consisting of a total of 18 statements such as "I understand", "I notice my special body reactions in case of extreme hunger". The participant will be asked to score for each statement from 1 (not at all true for me) to 7 (completely true for me). The total score in the questionnaire varies between 18-126, with higher scores indicating better body sensitivity (awareness).
Assessment of quality of life | 6 weeks
  Disease-related quality of life of young individuals included in the study, Alanay A. et al. It will be evaluated with the Scoliosis Research Society 22. Form (SRS 22r) scale, developed by the Scoliosis Research Society, which has been translated into Turkish and has proven validity and reliability. Scale "Which of the following answers best describes the pain you have experienced during the past 6 months?", "How much are you able to move now?", "How long have you felt calm and peaceful during the last 6 months?" It consists of 22 questions and 5 sub-dimensions. Sub dimensions; pain, self-image/view, spinal functions, mental health, and satisfaction with treatment. All of these sections are evaluated separately and/or all questions are collected under the total score. High scores indicate high quality of life
Assessment of pelvic shift | 6 weeks
  According to the C7-plumb line direction, considering the side where the central sacral vertical line is located, it will be recorded as "right and left shift" or "no shift" and pelvic asymmetry will be evaluated.
Assessment of Lower Extremity Length Measurement | 6 weeks
  The distance between the umbilicus and the medial malleolus will be measured in centimeters with a tape measure while the subjects are lying in the supine position. In some sources, it is stated that the measurement between spina illiaca anterior superior and medial malleolus is also used in lower extremity length measurements. In cases with scoliosis, measurement between the umbilicus and the medial malleolus will be preferred because there may be asymmetry in the pelvis.
Assessment of Pain | 6 weeks
  Visual Analogue Scale (VAS) will be used to evaluate the pain status of the patients. This scale, which is used to measure the severity of pain and has been validated and reliable, is a 10 cm line scaled from 1 to 10. A value of 10 indicates maximum pain, while a value of 0 means no pain. Individuals will be asked to mark a place on the scale according to the pain they feel at rest, during activity and at night, and the marked values will be recorded.
Assessment of Respiratory Muscles | 6 weeks
  It is planned to evaluate respiratory muscles by measuring maximal inspiratory (MIP) and expiratory (MEP) mouth pressure. MIP and MEP are parameters that show respiratory muscle strength and can be measured with portable small handheld devices. The device should contain a slight air leak to prevent the patient from generating additional pressure using the cheek muscles. MIP and MEP are measured using a flanged mouthpiece attached to a short, rigid tube with a three-way tap or valve system to ensure normal breathing followed by the MIP or MEP maneuver. The pressure in the tube is measured with a pressure transducer connected with a narrow calibrating catheter and the output from the strain gauge is displayed on the screen. The patient will be seated in an upright chair. He will be asked to grasp the silicone mouthpiece with his mouth and inhale and exhale as quickly and deeply as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- University of health sciences Istanbul physical therapy and rehabilitation training and research hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

REFERENCES:
- [Background] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Background] Rigo M, Reiter Ch, Weiss HR. Effect of conservative management on the prevalence of surgery in patients with adolescent idiopathic scoliosis. Pediatr Rehabil. 2003 Jul-Dec;6(3-4):209-14. doi: 10.1080/13638490310001642054. PMID 14713587